CLINICAL TRIAL: NCT03959449
Title: Action Observation and Motor Imagery Induced Hypoalgesia in Asymptomatic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: uammadrid8
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Analgesia; Exercise
Keywords: Motor imagery; Action observation; Hypoalgesia
MeSH Terms: conditions — Agnosia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action Observation and Motor imagery (Experimental)
  Interventions: Behavioral: Action Observation plus motor imagery
- Motor Imagery (Active Comparator)
  Interventions: Behavioral: Motor imagery
- Exercise plus motor imagery and action observation (Experimental)
  Interventions: Behavioral: Exercise plus action Observation and motor imagery

INTERVENTIONS:
Behavioral: Action Observation plus motor imagery — Action observation (video) and motor imagery of running.
  Arms: Action Observation and Motor imagery
Behavioral: Motor imagery — Motor imagery of running
  Arms: Motor Imagery
Behavioral: Exercise plus action Observation and motor imagery — Real exercise of running during 6 min plus action observation (video) and motor imagery of running.
  Arms: Exercise plus motor imagery and action observation

SUMMARY:
This study evaluates the influence of motor imagery and the observation of actions on pain perception. Participants in this study are asymptomatic subjects who will perform an IM and AO protocol of an aerobic exercise.

DETAILED DESCRIPTION:
Motor Imagery (MI) is defined as a dynamic mental process that involves the representation of an action, in an internal way, without its actual motor execution. The Action Observation (AO) evokes an internal, real-time motor simulation of the movements that the observer is perceiving visually. Both mental processes trigger the activation of the neurocognitive mechanisms that underlie the planning and execution of voluntary movements in a manner that resembles how the action is performed in a real manner. The phenomenon of exercise-induced hypoalgesia is well known. This is why it has been suggested that these techniques could produce pain modulation similar to that produced by real exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Healthy and with no pain subjects

Exclusion Criteria:

* Any cognitive impairment that hindered viewing of audiovisual material.
* Difficulty understanding or communicating.
* Presence of systemic pathology, Central Nervous System or rheumatic disease.
* Inadequate understanding of the Spanish language to follow instructions for measuring and treatment.
* Collaboration of pregnant women.
* Underage subjects
* Subjects with pain at the time of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Change from baseline and immediately post-intervention
  Pressure Pain Threshold (PPT) is one of these tests and it is defined as the minimum force applied which induces pain. The measurement shall be carried out by using an algometer (pressure device that induces mechanical stimuli) is to standardize the amount of pressure applied in the neck region. The reliability of pressure pain thresholds according to raters or measurement frequencies is relatively high

SECONDARY OUTCOMES:
Visual and Kinesthetic Motor Imagery Ability | Immediately before the intervention
  Visual and Kinesthetic Motor Imagery Ability will be measured with Movement Imagery Questionnaire-Revised (MIQ-R). MIQ-R has four movements repeated in two subscales, a visual and a kinesthetic one. Additionally, a score between 1 and 7 is assigned, with 1 representing difficulty in picturing the motor image or difficulty in feeling the movement previously made, and 7 representing the maximum ease. The internal consistencies of the MIQ-R have been consistently adequate with Cronbach's α coefficients ranging above 0.84 for the total scale, 0.80 for de visual subscale and 0.84 for the kinesthetic subscale (Campos & González, 2010).
The degree of physical activity | Immediately before the intervention
  The degree of physical activity was objectified through the The International Physical Activity Questionnaire (IPAQ) questionnaire, which allows the subjects to be divided into three groups according to their level of activity, which can be high, moderate, and low or inactive. The IPAQ consists of 7 questions about the frequency, duration and intensity of activity (moderate and intense) performed in the last seven days, as well as walking and sitting time on a workday. The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively.
Kinesiophobia | Immediately before the intervention
  Fear of movement or kinesiophobia will be quantified with the Spanish version of the Kinesiophobia Tampa Scale (TSK-11). This instrument demonstrates reliability and validity in patients with chronic pain, being shorter than the original scale. The total score ranges from 11 to 44 points, with the highest scores indicating greater fear of a new injury due to movement
Electrodermal Activity | Change in electrodermal activity after 5 minutes post-intervention
  Electrodermal Activity will be measured through the use of two electrodes that recorded changes in conductance through the skin located at the back of the dominant hand
Respiration Rate | Change in electrodermal activity after 5 minutes post-intervention
  Respiration Rate will be measured through a pressure transducer located in the centre of the chest, where it was fixed by a strap
Respiration Rate | Change in electrodermal activity after 5 minutes post-intervention
  Heart Rate will be measured by three electrodes located in the left area of the chest. One of the electrodes was placed in the middle zone while a second electrode was positioned on the lateral side, and a third one on the lower left side, below the first electrode.

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No